CLINICAL TRIAL: NCT05553509
Title: Clinical Outcomes Following Surgical Debridement of Diabetic Foot Infection with Borderline Vascularity: an Important Consideration of Timing of Revascularization
Brief Title: Clinical Outcomes Following Surgical Debridement of Diabetic Foot Infection with Borderline Vascularity
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Ayman Hussien Shaamash, Principal investigator, Assiut University
Other Study IDs: AST-KASH-ENDO
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Limb Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ANGIOPLASTY GROUP: All patients undergoing PTA are going to be classified according to GLASS staging system
  Interventions: Other: PER CUTANEOUS TRANSLUMINAL ANGIOPLASTY
- DEBRIDEMENT GROUP: The most commonly used technique for diabetic foot ulcers is sharp or surgical debridement using a scalpel, tissue forceps or similar instruments. It should be sufficiently extensive to remove all infected and necrotic tissue;
  Interventions: Other: PER CUTANEOUS TRANSLUMINAL ANGIOPLASTY

INTERVENTIONS:
Other: PER CUTANEOUS TRANSLUMINAL ANGIOPLASTY — SURGICAL DEBRIDEMNT
  Other Names: REVASCULARIZATION

SUMMARY:
Observe Timing to complete healing of wounds & Limb salvage in both cohorts those who are undergoing Debridement only and those who are undergoing Debridement plus PTA

DETAILED DESCRIPTION:
Secondary Aims of the study include Length of hospital stay , Necessity of further intervention(Whether a Revascularization Procedure or More Debridement sessions) , Incidence of MACE (Major Adverse Cardiovascular Events) in both groups

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in this study are those suffering from DFUs; and Borderline Ischemia (BLI) / Borderline Vacularity with (Rutherford Grade "I" Categories "2&3") when they have a borderline ankle systolic pressure

Exclusion Criteria:

* All patients with (CLI) and DFUs as they are indicated for urgent re-vascularization.

Severely infected/ gangrenous wounds requiring amputation hindering possible limb salvage.

Lesions lying within or adjacent to an aneurysm; Non diabetic cases with foot ulcers; Arteritic lesions;(Vasculitic Patients). Patients had prior major amputation, bypass surgery, and endarterectomy on any vessel of the ipsilateral (target) extremity

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: On the other hand we can consider patients as Borderline ischemia/ Boarderline Vascularity with (Rutherford Grade "I" Categories "2&3) when they have a borderline ankle systolic pressure
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes Following Surgical Debridement of Diabetic Foot Infection With Borderline Vascularity | 1 YEAR
  1. Observe the timing to complete wound healing in both cohorts those with Debridement only & those with Debridment plus PTA
  2. Observe the Rate of limb salvage in both groups

SECONDARY OUTCOMES:
Clinical Outcomes Following Surgical Debridement of Diabetic Foot Infection With Borderline Vascularity | 1 YEAR
  1-Observe incidence of MACE In both cohorts Observe necessity for further interventions in both cohorts 3-Observe the length of hospital stay in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of vascular surgery - Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No